CLINICAL TRIAL: NCT02957721
Title: DEAP: Diabetes Engagement and Activation Platform
Brief Title: Diabetes Engagement and Activation Platform
Acronym: DEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM20008890
Record Dates: First submitted 2016-10-28; First posted 2016-11-08 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes (T2D)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral self-management (Other): Eligible patients who are registered on the practice EHR linked portal will be invited to join the study. Following informed consent, enrollment and randomization, participants in the treatment group will receive the type 2 diabetes behavioral self-management education intervention; comprised of 9 modules derived from Medline Plus.
  Interventions: Other: Usual Care
- Usual Care (No Intervention): Usual care includes whatever care and services the patient's clinical provides as well as generic type 2 diabetes education built into the patient's EHR linked portal.

INTERVENTIONS:
Other: Usual Care — Patients will not be given the intervention but receive usual care for T2D.
  Arms: Behavioral self-management

SUMMARY:
The following are hypothesized:

1. The Diabetes Engagement and Activation Platform (DEAP) can be integrated into primary care workflow to facilitate the care of patients with type 2 diabetes.
2. The DEAP intervention will be feasible and acceptable to patients with type 2 diabetes.
3. The DEAP intervention will enhance patient activation and improve type 2 diabetes self management and glucose control

DETAILED DESCRIPTION:
Aim 1: To evaluate how primary care practices adopt and integrate DEAP into routine workflow including identification of barriers and facilitators to support acceptable, feasible, and sustainable use of the system.

* Sub-aim 1.1: Measure the proportion of clinicians and care team members who engage patients through the DEAP intervention as well as the types of patient support activities they address; assess the representativeness of participating clinicians and care team members in relation to all practice staff; and assess how they integrated DEAP into the care of type 2 diabetes patients.
* Sub-aim 1.2: Assess how practices redesign workflow, overcome barriers, and enhance facilitators in order to integrate DEAP.
* Sub-aim 1.3: Determine processes for sustaining DEAP beyond the project funding period .

Aim 2: To compare, relative to usual care, the effectiveness of the DEAP intervention.

* Sub Aim 2.1: Measure the proportion and representativeness of eligible patients who choose to enroll; access the DEAP curriculum; complete the DEAP curriculum; and contact care team members. .
* Sub Aim 2.2: Compare the change in the average glycosylated hemoglobin (primary outcome), Body Mass Index, systolic blood pressure, and type 2 diabetes (T2D) medications and patient activation (secondary outcomes) from baseline to 3 months and from 3 to 6 months for patients randomized to DEAP versus usual care.

Sub Aim 2.3: Assess the clarity, readability and acceptability of the DEAP curricula materials for T2D patients enrolled in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes and A1C measure ≥ 8%;
* English speaking;
* Enrolled in the practice EHR linked patient portal.

Exclusion Criteria:

* Patients without type 2 diabetes or with type 2 diabetes who have a A1C less than or equal to 7.9%;
* Non-English speaking;
* Patients not enrolled in the practice EHR linked patient portal;
* Under 18 and over 75 years of age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Change in A1C | From date of study enrollment A1C will be retrieved from electronic health record (EHR) at baseline, 3 and 6 months after enrollment. Data will continue to be collected at these intervals on all participants until target sample of 160 is complete.
  The A1C test is a blood test that provides information about a person's average levels of blood glucose, also called blood sugar, over the past 3 months. The A1C test is sometimes called the hemoglobin A1c, HbA1c, or glycohemoglobin test.

SECONDARY OUTCOMES:
Patient Activation Measure (PAM 10) | From date of study enrollment PAM 10 will be retrieved from patient portal at baseline, 3 and 6 months following enrollment. Data will continue to be collected at these intervals on all participants until target sample of 160 is complete.
  measures how well patients self-manage diabetes.
Body Mass Index (BMI) | From date of study enrollment BMI will be retrieved from EHR at baseline, three and six months following enrollment. Data will continue to be collected at these intervals on all participants until target sample of 160 is complet
  The BMI is an attempt to quantify the amount of tissue mass (muscle, fat, and bone) in an individual, and then categorize that person as underweight, normal weight, overweight, or obese based on that value.
Blood Pressure (BP) | From date of study enrollment BP will be retrieved from EHR at baseline, 3 and 6 months following enrollment. Data will continue to be collected at these intervals on all participants until target sample of 160 is complete.
  Systolic blood pressure represents the pressure in the arteries when the heart is contracting, and the pressure when the heart is at rest is called diastolic blood pressure. Blood pressure is measured using a blood pressure cuff, which is wrapped around the upper arm.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander H Krist, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sabo R, Robins J, Lutz S, Kashiri P, Day T, Webel B, Krist A. Diabetes Engagement and Activation Platform for Implementation and Effectiveness of Automated Virtual Type 2 Diabetes Self-Management Education: Randomized Controlled Trial. JMIR Diabetes. 2021 Mar 29;6(1):e26621. doi: 10.2196/26621. PMID 33779567